CLINICAL TRIAL: NCT03502512
Title: A Randomized, Prospective Comparison of Methods to Process Autologous Fat Grafts in Breast Reconstruction
Brief Title: REVOLVE or PureGraft Technique in Processing Fat Grafts for Patients Undergoing Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0463; NCI-2018-00944 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0463 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Mammoplasty Patient
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (REVOLVE technique) (Experimental): Patients undergo reconstructive surgery with REVOLVE technique.
  Interventions: Other: Questionnaire Administration; Procedure: Reconstructive Surgery
- Arm II (PureGraft technique) (Experimental): Patients undergo reconstructive surgery with PureGraft technique.
  Interventions: Other: Questionnaire Administration; Procedure: Reconstructive Surgery

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Procedure: Reconstructive Surgery — Undergo reconstructive surgery with REVOLVE technique
  Other Names: Reconstruction
  Arms: Arm I (REVOLVE technique)
Procedure: Reconstructive Surgery — Undergo reconstructive surgery with PureGraft technique
  Other Names: Reconstruction
  Arms: Arm II (PureGraft technique)

SUMMARY:
This trial studies how well REVOLVE or PureGraft technique works in processing fat grafts for patients who are undergoing breast reconstruction. During breast reconstructive surgery that uses autologous fat grafting (transplanting fat tissue from one part of your body to another), fat tissue is removed from the body (usually the abdomen, buttock, or thighs) and injected into another part of the body. This tissue must be "processed" (sometimes referred to as "washed" or "prepared") before being inserted back into the body. It is not yet known whether REVOLVE or PureGraft technique may work better in retaining graft fat after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure and compare the rate of fat graft retention, defined as the rate between the volume of fat remaining in the surgical site at one year and the volume of fat at baseline, associated with the use of two aforementioned adipose tissue processing techniques.

SECONDARY OBJECTIVES:

I. To measure early post-operative complications including infection, hematoma, delayed wound healing or seroma.

II. To measure late complications associated with fat grafting including fat necrosis, cyst formation, palpable mass, or breast asymmetry.

III. To measure patient reported outcomes (PRO, BREAST-Questionnaire [Q], Body Image Survey).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo reconstructive surgery with REVOLVE technique.

ARM II: Patients undergo reconstructive surgery with PureGraft technique.

After completion of study, patients are followed up at 2-4 weeks and then once a year for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Previous breast surgery, either mastectomy or partial mastectomy
* Patients with available harvest sites for fat grafting
* Patients with body mass index (BMI) > 20
* Anticipated harvested fat volume > 100 cc
* Patients are willing and able to give consent

Exclusion Criteria:

* Patients with active cancer, including primary cancer, recurrent cancer and locally or distantly metastatic cancer
* Patients who are unable to provide consent
* Patients who are suspected or known to be pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Fat graft retention rate | At 1 year
  Rate of fat graft retention, defined as the rate between the volume of fat remaining in the surgical site at one year and the volume of fat at baseline, associated with the use of the REVOLVE and PureGraft tissue processing techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reece, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org